CLINICAL TRIAL: NCT04269772
Title: Project CARE (Community Treatment Adherence at Re-Entry): An Integrated Treatment Adherence Program for Bipolar Disorder at the Time of Prison Release - Pilot RCT
Brief Title: Project CARE: An Integrated Treatment Adherence Program for Bipolar Disorder at the Time of Prison Release - Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1806002090-RCT; R34MH117198 (NIH)
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2023-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community treatment Adherence at Re-Entry (CARE) (Experimental): CARE will begin within the 2 months before prison release, and will continue for 6 months after re-entry. CARE will be comprised of: a) 3 individual sessions with the CARE counselor; b) 1 optional family/significant other (SO) session; and c) 11 brief (15-20 min) follow-up telephone contacts with prisoners and their SO over the first 6 months post-release.
  The CARE intervention will incorporate motivational strategies from existing interventions (e.g., Acceptance and Commitment Therapy) in order to clarify values and goals to enhance motivation for community treatment engagement and behavior change. CARE will also integrate bipolar disorder psychoeducation and strategies from existing models of intervention for BD (e.g., McMaster Model of Family Functioning) that are designed to improve family communication, social support, and problem-solving around BD illness management over this vulnerable transition period.
  Interventions: Behavioral: CARE
- Treatment As Usual (TAU) (Other): Treatment As Usual (TAU) consists of unrestricted treatment provided by prison and community providers, as part of routine care in the criminal justice re-entry context. Study staff will provide no additional treatment in this arm.
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Behavioral: CARE — Hybrid in-person and telephone-based adjunctive intervention for bipolar disorder across the transition from prison to the community.
  Arms: Community treatment Adherence at Re-Entry (CARE)
Other: Treatment As Usual — Treatment as usual, unrestricted, as provided by prison and community providers.
  Arms: Treatment As Usual (TAU)

SUMMARY:
The aim of this program of research is to develop and pilot the CARE (Community treatment Adherence at Re-Entry) program, an adjunctive intervention for incarcerated individuals with bipolar disorder (BD) transitioning from prison to the community.

The purpose of this proposed project is to establish the feasibility, acceptability, and preliminary effects of this newly developed intervention on symptom outcomes in a small pilot randomized controlled feasibility trial.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a serious, disabling, and highly recurrent illness that is disproportionately represented in the criminal justice system. BD increases risk for several adverse outcomes for prisoners, including mood instability, suicide attempts, substance use relapse, and high rates of repeat incarceration. Despite these serious negative consequences, up to 70% of prisoners with BD do not receive mental health treatment upon prison release. Lack of engagement in ongoing mental health treatment for BD upon community re-entry represents one potent factor that perpetuates risk for adverse outcomes, and consequences of untreated BD (e.g., impulsivity, substance use) may greatly exacerbate difficulties in establishing stable living conditions (e.g., adequate housing, legal employment) at community re-entry. Thus, there is a critical need for interventions to facilitate engagement with treatment for BD during this vulnerable transition.

To that end, the primary aim of this study is to develop and establish the feasibility and acceptability of the Community treatment Adherence at Re-Entry (CARE) program. CARE is an innovative intervention that will combine evidence-based cognitive-behavioral, family, and telephone outreach strategies to promote treatment engagement and improve clinical outcomes for prisoners with BD during the period of community re-entry. CARE will include 3 individual and 1 family session, followed by 11 brief telephone contacts for up to 6 months post-release. Given its moderate intensity, adjunctive nature, use of community mental health counselors, and use of telephone administration of post-release follow-up, CARE has been designed with an eye toward community implementation. Its proposed mechanisms of action (i.e., increasing values-action consistency, enhancing social supports, and linkage to community treatment services) are further well matched to the practical and clinical needs of re-entering individuals.

The aim of this research is to conduct a small pilot randomized controlled trial (n=40) of the CARE intervention compared to treatment as usual for prisoners with BD around the time of community re-entry. Assessments will occur at baseline, immediately pre-release, 4 weeks post-release, and 24 weeks post-release (post-treatment). This study will examine the feasibility and acceptability of CARE (e.g., update, adherence to, and completion of the CARE intervention, satisfaction with the intervention, understanding of intervention principles) and of this research design. This study will also examine treatment effects (within relevant confidence intervals) on outcomes (e.g., mood symptoms). Change in potential mechanisms (i.e., values-action consistency derived from intervention principles) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of bipolar I, bipolar II, or bipolar disorder not elsewhere classified
* Anticipated prison release within 4-10 weeks
* Expected release to locations anywhere in RI or to locations in other states within a 30 mile radius of Providence
* Aged 18 or older
* Willingness to sign an informed consent document that describes study procedures

Exclusion Criteria:

* Presence of current psychiatric symptoms severe enough to warrant separation from the general prison population
* Cognitive impairment sufficient to prevent successful completion of the baseline interview
* Inability to understand English sufficiently well to understand the consent form or assessment instruments when they are read aloud

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Weinstock, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Department of Corrections, Cranston, Rhode Island
  - Brown University, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Treatment Adherence at Re-Entry (CARE): CARE will begin within the 2 months before prison release, and will continue for 6 months after re-entry. CARE will be comprised of: a) 3 individual sessions with the CARE counselor; b) 1 optional family/significant other (SO) session; and c) 11 brief (15-20 min) follow-up telephone contacts with prisoners and their SO over the first 6 months post-release.
  The CARE intervention will incorporate motivational strategies from existing interventions (e.g., Acceptance and Commitment Therapy) in order to clarify values and goals to enhance motivation for community treatment engagement and behavior change. CARE will also integrate bipolar disorder psychoeducation and strategies from existing models of intervention for BD (e.g., McMaster Model of Family Functioning) that are designed to improve family communication, social support, and problem-solving around BD illness management over this vulnerable transition period.
  CARE: Hybrid in-person and telephone-based adjunctive intervention for bipolar disorder across the transition from prison to the community.
- Significant Others (SOs): Significant Others (SOs) are enrolled to support the participant in their study treatment (CARE). SOs only participate in family sessions and brief phone sessions (as described in the CARE arm). SO enrollment is optional.
Period: Overall Study
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU) | Significant Others (SOs)
Started | 15 | 15 | 4
Completed | 14 | 15 | 4
Not Completed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU) | Significant Others (SOs) | Total
Number analyzed (Participants) | 15 | 15 | 4 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.07 (9.45) | 37.00 (9.99) | 44.25 (17.75) | 37.44 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 4 | 14
  Male | 10 | 10 | 0 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 12 | 14 | 3 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 7 | 10 | 2 | 19
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 4 | 34

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire-8 (CSQ-8)
Description: Intervention feasibility and acceptability. Total Client Satisfaction Questionnaire-8 (CSQ-8) scores range from 8 to 32 with higher scores indicating higher levels of satisfaction.
Time Frame: 24 weeks post-release
Population: Note: Out of the 14 participants that completed the study in the CARE arm, only 8 completed the CSQ-8 at the 24 week follow-up (6 did not complete it). Out of the 15 participants that completed the TAU arm, only 10 completed the CSQ-8 at the 24 week follow-up (5 did not complete it). Additionally, Outcome Measure data was not collected for SOs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU)
Number analyzed (Participants) | 8 | 10
score on a scale | 28.00 (6.57) | 26.20 (5.16)

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR)
Description: Depressive symptom severity. Total QIDS-SR depressive symptom severity scores range from 0 to 27 with higher scores indicating more severe depressive symptoms.
Time Frame: 24 weeks post-release
Population: Note: Out of the 14 participants that completed the study in the CARE arm, only 8 completed the QIDS-SR at the 24 week follow-up (6 did not complete it). Out of the 15 participants that completed the TAU arm, only 11 completed the QIDS-SR at the 24 week follow-up (4 did not complete it). Additionally, Outcome Measure data was not collected for SOs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU)
Number analyzed (Participants) | 8 | 11
score on a scale | 7.38 (6.61) | 7.64 (5.82)

3. Secondary Outcome: Altman Self-Rating Scale for Mania (ASRM)
Description: Manic symptom severity. Total Altman Self-Rating Scale for Mania (ASRM) manic symptom severity scores range from 0 to 20 with higher scores indicating more severe symptoms of mania.
Time Frame: 24 weeks post-release
Population: Note: Out of the 14 participants that completed the study in the CARE arm, only 8 completed the ASRM at the 24 week follow-up (6 did not complete it). Out of the 15 participants that completed the TAU arm, only 11 completed the ASRM at the 24 week follow-up (4 did not complete it). Additionally, Outcome Measure data was not collected for SOs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU)
Number analyzed (Participants) | 8 | 11
score on a scale | 1.13 (2.10) | 1.82 (2.44)

ADVERSE EVENTS:
Time Frame: Assessed from consent through 24 weeks post-release, up to 38 weeks
Description: Adverse Event data was only collected from the main study participants. It was not collected from SOs.
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15 | 1/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community Treatment Adherence at Re-Entry (CARE) (N=15) | Treatment As Usual (TAU) (N=15)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) — Non-fatal suicide attempt
Inpatient Hopsitalization (Psychiatric disorders) | 1 (1) | 1 (1) — Suicide or potentially suicide related inpatient hospitalization

LIMITATIONS AND CAVEATS:
Recruitment began 01/20/20 but was paused 03/12/20 due to COVID-related prison lockdowns. In consultation w/ RIDOC admin and Brown University IRB, an additional recruitment method was approved in which the prison provided referrals of individuals just released from prison, for approach by phone for post-release study enrollment; referral-based recruitment began 10/05/20.The study received permission to resume in-person recruitment in the prison on 09/18/21, per the original recruitment protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT04269772/Prot_SAP_000.pdf